CLINICAL TRIAL: NCT02132533
Title: Nifedipine for Acute Tocolysis of Preterm Labor
Acronym: Nifedipine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 122013-063
Record Dates: First submitted 2014-04-30; First posted 2014-05-07 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nifedipine (Experimental): Women with preterm labor will receive nifedipine.
  Interventions: Drug: Nifedipine; Other: Usual care
- Placebo (Experimental): Women with preterm labor will receive placebo.
  Interventions: Drug: Placebo; Other: Usual care

INTERVENTIONS:
Drug: Nifedipine — Nifedipine 20 mg orally, then nifedipine 20 mg orally after 90 minutes if still contracting. Continue nifedipine 20 mg orally every 4 hours after the first dose for 48 hours.
  Arms: Nifedipine
Drug: Placebo — Placebo orally, then placebo orally after 90 minutes if still contracting. Continue placebo orally every 4 hours after the first dose for 48 hours.
  Arms: Placebo
Other: Usual care — Usual evaluation, monitoring and care for women with preterm labor.

SUMMARY:
The purpose of this study is to determine if nifedipine treatment of women in preterm labor receiving corticosteroids results in postponement of delivery when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Between 16 and 44 years of age inclusive
* Singleton pregnancy
* Intact membranes
* Between 28-0/7 weeks and 33-6/7 weeks' gestation inclusive
* Reported or documented uterine activity
* Cervical dilation between 2 cm and 4 cm inclusive

Exclusion Criteria:

* Multifetal gestation
* Less than 28 weeks' gestation
* 34 or more weeks' gestation
* Ruptured membranes
* More than 4 cm dilated
* Previously received a course of corticosteroids for fetal lung maturation
* Oligohydramnios
* Fetal growth restriction
* Chorioamnionitis or temperature of at least 38.0 degrees Celsius
* Fetal death
* Preeclampsia
* Suspected placental abruption or placenta previa
* Lethal fetal malformation or amniotic fluid index at least 35
* Systolic BP < 90 mmHg or diastolic BP < 50 mmHg
* Baseline tachycardia (pulse >120 after 2 consecutive measurements 30 minutes apart)
* Chronic hypertension treated with antihypertensives in pregnancy
* Seizure disorder or HIV
* Maternal allergy to nifedipine
* Known maternal cardiac disease
* Women who have received progesterone therapy in the second or third trimester for prevention of preterm birth

Ages: 16 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2014-05-05 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Casey, MD, Study Director — Department of Alabama Medical Center, Birmingham, AL; Donald D McIntire, PhD, Study Director — University of Texas Southwestern Medical Center; Kenneth J Leveno, MD, Study Director — University of Texas Southwestern Medical Center; Chet E Wells, MD, Study Director — University of Texas Southwestern Medical Center; Josiah S Hawkins, MD, Principal Investigator — Kaiser Medical Center, Oakland, CA
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046
- [Derived] Hawkins JS, Wells CE, Casey BM, McIntire DD, Leveno KJ. Nifedipine for Acute Tocolysis of Preterm Labor: A Placebo-Controlled Randomized Trial. Obstet Gynecol. 2021 Jul 1;138(1):73-78. doi: 10.1097/AOG.0000000000004436. PMID 34259466

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nifedipine | Placebo
Started | 46 | 42
Completed | 46 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nifedipine | Placebo | Total
Number analyzed (Participants) | 46 | 42 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 5 | 6
  Between 18 and 65 years | 45 | 37 | 82
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (5.8) | 26.7 (6.7) | 26.1 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 42 | 88
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 10 | 6 | 16
  White | 1 | 1 | 2
  Hispanic | 35 | 35 | 70
Region of Enrollment [Number; unit: participants]
  United States | 46 | 42 | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Preterm Birth
Time Frame: Less than 37 weeks of gestation
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Placebo
Number analyzed (Participants) | 46 | 42
Participants | 24 | 20

2. Secondary Outcome: Number of Participants With Preterm Birth
Time Frame: Within 48 hours of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Placebo
Number analyzed (Participants) | 46 | 42
Participants | 8 | 10

3. Secondary Outcome: Number of Participants With Preterm Birth
Time Frame: At least 2 doses of betamethasone administered prior to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Placebo
Number analyzed (Participants) | 46 | 42
Participants | 36 | 31

4. Secondary Outcome: Number of Participants With Preterm Birth
Time Frame: Within 7 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Placebo
Number analyzed (Participants) | 46 | 42
Participants | 13 | 14

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Nifedipine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/42
Other Adverse Events (participants affected / at risk) | 0/46 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT02132533/Prot_SAP_000.pdf